CLINICAL TRIAL: NCT04806568
Title: Cognitive Decline Prognosis in Multiple Sclerosis: Effectiveness of a Computerized Cognitive Training Treatment on Cortical Reorganization
Brief Title: MS-NEUROPLAST: Neuroplasticity of Cortical Areas Induced by Cognitive Training in Patients with Multiple Sclerosis
Acronym: MSNEUROPLAST
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Aristotle University Of Thessaloniki (Other)
Collaborators: King Fahad Medical City (Other Government)
Responsible Party: Principal Investigator, Panos Bamidis, Professor, Aristotle University Of Thessaloniki
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 98223
Record Dates: First submitted 2021-03-03; First posted 2021-03-19 (Actual); Last update posted 2024-11-04 (Actual); Status verified 2024-10

CONDITIONS: Multiple Sclerosis; Cognitive Decline
Keywords: EEG; Network Efficiency; Adaptive; Plasticity; Maladaptive Reorganization; Cognitive Training
MeSH Terms: conditions — Multiple Sclerosis; Cognitive Dysfunction | interventions — Cognitive Training

STUDY DESIGN:
Intervention Model Description: Patients will wear a smartwatch and will be randomly assigned to either the cognitive intervention, or the active control group, stratified by age, sex, education and cognition.
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- PwMS-CCT (Experimental): Adult individuals with Multiple Sclerosis will follow a cognitive training intervention.
  * Neurological assessment
    * History of Multiple Sclerosis
    * Expanded Disability Status Scale (EDSS)
  * 2 types of high-density electroencephalographic recordings
    * at rest with eyes closed (15 minutes)
    * event potentials via a multisensory oddball paradigm (45 minutes)
  * Neuropsychological assessment
    * MMSE
    * CDT
    * GVLT
    * BVMT
    * SDMT
    * Verbal Fluency: Phonemic [ Chi-Sigma-Alpha] and Semantic [Animals-Fruits-Objects]
    * Digit Span (For-Back-Seq)_WAIS-4GR
    * SNST
    * GAT
    * DASS21
    * MSIS-29
    * CRIq
    * MFIS
    * EQ-5D-5L
    * BDI-II
  * Somatometric assessment
    * Timed 25-Foot Walk (T25-FW)
    * 3m backwards walk test
    * Hole Peg Test (9-HPT)
    * Handgrip Strength Test
    * Single Leg Stance (SLS)
    * Four Square Step Test (FSST)
  * BrainHQ training
  * Monitoring of daily activity
  Interventions: Other: Cognitive Training; Device: Monitoring of daily activity
- PwMS-CON (Active Comparator): Adult individuals with Multiple Sclerosis serving as active controls.
  * Neurological assessment
    * History of Multiple Sclerosis
    * Expanded Disability Status Scale (EDSS)
  * 2 types of high-density electroencephalographic recordings
    * at rest with eyes closed (15 minutes)
    * event potentials via a multisensory oddball paradigm (45 minutes)
  * Neuropsychological assessment
    * Mini Mental Status Examination (MMSE)
    * Clock Drawing Test (CDT)
    * Greek Verbal Learning Test (GVLT)
    * Brief Visuospatial Memory Test (BVMT)
    * Symbol Digit Modalities Test (SDMT)
    * Verbal Fluency: Phonemic [ Chi-Sigma-Alpha] and Semantic [Animals-Fruits-Objects]
    * Digit Span (For-Back-Seq)_WAIS-4GR
    * Stroop Neuropsychological Test (SNST)
    * The Greek Accentuation Test (GAT)
    * DASS-21
    * MSIS-29
    * CRIq
    * MFIS
    * EQ-5D-5L
    * BDI-II
  * Somatometric assessment
    * T25-FW
    * 3m backwards walk test
    * 9-HPT
    * Handgrip Strength Test
    * SLS
    * FSST
  * Monitoring of dailty activity
  Interventions: Device: Monitoring of daily activity
- HC (No Intervention): Healthy adults serving as passive controls.
  * 2 types of high-density electroencephalographic recordings
    * at rest with eyes closed (15 minutes)
    * event potentials via a multisensory oddball paradigm (45 minutes)
  * Neuropsychological assessment
    * Mini Mental Status Examination (MMSE)
    * Greek Verbal Learning Test (GVLT)
    * Brief Visuospatial Memory Test (BVMT)
    * Symbol Digit Modalities Test (SDMT)
  * Somatometric assessment
    * Timed 25-Foot Walk (T25-FW)
    * 3m backwards walk test
    * Hole Peg Test (9-HPT)
    * Handgrip Strength Test
    * Single Leg Stance (SLS)
    * Four Square Step Test (FSST)

INTERVENTIONS:
Other: Cognitive Training — The cognitive training treatment is a Greek adaptation of BrainHQ developed by Posit Science Corporation. The intervention will target speed, attention, working memory, and executive function through the visual and auditory domains via a set of 15 exercises. Each daily training session consists of four exercises chosen from an active set of six. Participants will be instructed to train for one hour per day, three days per week, over 12 weeks via a tablet. Each subject will receive at least 29 sessions of computerized cognitive training.
  Arms: PwMS-CCT
Device: Monitoring of daily activity — Monitoring of daily activity via Fitbit Charge 4 smartwatch.
  Arms: PwMS-CCT; PwMS-CON

SUMMARY:
This clinical study aims to identify MS related beneficial plasticity and by contrast maladaptive reorganization in combination with elements of daily functional status as a response to a cognitive training program

DETAILED DESCRIPTION:
Cognitive decline is a debilitating and widespread comorbidity of Multiple Sclerosis (MS) affecting up to 65 percent of patients with MS (PwMS). Cognitive changes can be the only behavioral index of MS activity. But how accurately and timely can these be captured? The existing clinical tools are subjective and do not have the dynamic of prognosis. It remains uncertain how much change in cognitive status is required to translate into a meaningful clinical outcome and how long it may subsequently take to become apparent. Moving towards a holistic approach, MS-NEUROPLAST aims to further expand previously-published prognostic marker candidates and previous work of the applicant and the members of the research team and employ a group of methodologies for interventions and applications which will quantify via real-world assessment the MS-related cognitive changes in order to characterize not only decline but given the right dosage of stimulation improvement as well.

MS-NEUROPLAST has three main objectives:

(i) Utilize state of-the-art neuroimaging and network science measures to more thoroughly understand neural indices of cognitive impairment in PwMS.

(ii) Evaluate the efficacy for treating MS-associated cognitive deficits using a computerized cognitive training treatment by determining the differences, between subjects treated with cognitive training and controls, on network science measures indexing network efficiency or collapse and on the performance of a battery of neuropsychological tests that are frequently impaired in MS.

(iii) Investigate the dissociation of the cortical mechanisms related to training-induced plasticity and maladaptive reorganization (namely separate good from bad), by taking into account the homeostatic capacity of the human organism as a whole and thus examining whether the correlation of the neurophysiological and cognitive indices with longitudinal digital biomarkers of daily functional status can capture the underlying pathology.

MS-NEUROPLAST stages for PwMS

1. Provide signed informed consent to participate in the study after being informed by the principal investigator.
2. Neurological evaluation and decision on whether the inclusion criteria are met.
3. The participants will visit the Medical Physics & Digital Innovation Lab at AUTH, where:

   A. They will undergo a neuropsychological and somatometric assessment

   B. Then, they will undergo an electroencephalogram (EEG) measurement which includes the following:
   * Placement of the EEG cap holding the electrodes on the head to record the electrical activity of the brain. The cap will be soaked with potassium chloride solution to maintain the electrodes' resistance at desired levels
   * Wear over ear headphones
   * Recording EEG activity at rest for 15 minutes with eyes closed
   * View and listen to a series of simple images and sounds in video format and parallel recording of EEG evoked potentials using a complex eccentric (oddball) protocol combining multisensory audiovisual mismatches with unisensory acoustic and visual deviancies. Concurrently to the EEG measurements the subjects will respond behaviourally via button presses to an audiovisual congruency task on which they have to evaluate whether the images presented correspond to the tones they hear based on the rule: "the higher the pitch of the tone the higher the position of the circle". The recording will be performed 4 times, will include 32 sequences from each category audiovisual congruent, audiovisual incongruent, auditory deviant and visual deviant) resulting in 128 measurements from each condition for each participant. The measurement will take about 45 minutes.

   C. Familiarization with using a personal computer or a tablet, and demonstration of both the BrainHQ environment for cognitive training and the wearable and ambient devices.
4. Use of a set of smart sensors to collect biomarkers (steps, calories, sleep duration, heart rate, oxygen saturation) of daily activities for a period of up to 1 month (at least 2 weeks) before the onset of cognitive training. This will be followed by cognitive training through BrainHQ exercises. The training should be performed with a frequency of at least 3 times a week, for about 60 minutes (30 minutes of pure practice), lasting up to 12 weeks. Adherence will be recorded by the BrainHQ application and any deviations from the schedule will be followed by communication via the telephone or in person aimed at mobilizing and re engaging participants. During cognitive training, the recording of biomarkers of daily activities will continue.
5. At the end of the training, stages 3A and 3B will be repeated.

MS-NEUROPLAST stages for Healthy Controls

1. Provide signed informed consent to participate in the study after being informed by the principal investigator
2. The participants will visit the Medical Physics & Digital Innovation Lab at AUTH, where:

A. They will undergo a neuropsychological and somatometric assessment

B. Then, they will undergo an electroencephalogram (EEG) measurement which includes the following:

* Placement of the EEG cap holding the electrodes on the head to record the electrical activity of the brain. The cap will be soaked with potassium chloride solution to maintain the electrodes' resistance at desired levels
* Wear over ear headphones
* Recording EEG activity at rest for 15 minutes with eyes closed
* View and listen to a series of simple images and sounds in video format and parallel recording of EEG evoked potentials using a complex eccentric (oddball) protocol combining multisensory audiovisual mismatches with unisensory acoustic and visual deviancies. Concurrently to the EEG measurements the subjects will respond behaviourally via button presses to an audiovisual congruency task on which they have to evaluate whether the images presented correspond to the tones they hear based on the rule: "the higher the pitch of the tone the higher the position of the circle". The recording will be performed 4 times, will include 32 sequences from each category audiovisual congruent, audiovisual incongruent, auditory deviant and visual deviant) resulting in 128 measurements from each condition for each participant. The measurement will take about 45 minutes.

ELIGIBILITY:
Inclusion Criteria for people with MS:

* Male/female patients aged 18 to 65 years at screening
* Diagnosis of MS according to the 2017 Revised McDonald criteria
* Disability status at screening with an EDSS score of 0 to 6.5
* Relapsing MS and progressive MS as defined by Lublin
* Neurologically stable within 1 month prior to screening
* Patients receiving the same Disease Modifying Treatment (DMT) for at least 6 months

Exclusion Criteria for people with MS:

* Patients suspected of not being able or willing to cooperate or comply with study protocol requirements
* Patients meeting criteria for other demyelinating diseases of the CNS
* Patients with active chronic disease (or stable but treated with immune therapy) of the immune system other than MS
* Patients with any other significant CNS disease or serious psychiatric disorder which can interfere with the patient's ability to cooperate or comply with the study procedure
* Patients unable or unwilling to undergo MRI scans and EEG

Inclusion Criteria for Healthy Controls:

• Normal hearing and normal or corrected-to-normal vision

Exclusion Criteria for Healthy Controls:

* Any diagnosed neurological, mental, developmental, or psychiatric disorder
* Unrecovered neurological disorders (i.e., stroke, traumatic brain injury)
* Unstable medication within the last 3 months
* Intake of central nervous drugs (e.g., antidepressants)
* Severe physical disorder
* Concurrent participation in another relevant study
* Patients unable or unwilling to undergo EEG measurements

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 180 (Estimated)
Dates: Start 2020-12-01 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Change in current density strength of the cortical activity as measured via EEG | 3 months
  Changes in cortical activity strength caused via the training. Change is defined as statistical significance in the t-test comparison of the current density strength as reconstructed via Low Resolution Electromagnetic Tomography (LORETA) algorithm on the basis of high-density EEG recordings, before compared to after the training.
Change in cortical connectivity as measured via EEG | 3 months
  Changes in cortical connectivity caused via the training. Change is defined as statistical significance in the t-test comparison of Phase Transfer Entropy estimated from the cortical activity, as reconstructed via LORETA algorithm on the basis of high density EEG recordings, before compared to after the training.
Changes in the graph theory indexes as measured via EEG | 3 months
  Changes in the global and local graph theoretical indices of the brain networks caused via the training. Change is defined as statistical significance in the t-test comparison of the graph theory indices before compared to after the training.

SECONDARY OUTCOMES:
Change in audiovisual integration functionality | 3 months
  Change of accuracy in the behavioral measurement testing audiovisual integration. Change is defined as statistical significance in the t-test comparison before compared to after the training. A lower score denotes a decline.
Change in Mini Mental Status Examination (MMSE) | 3 months
  The Mini-Mental State Exam (MMSE) is a test of cognitive function. It includes tests of orientation, attention, memory, language, and visual-spatial skills.
  Change is defined as statistical significance in the comparison between before and after the training.
  The score ranges from 0 (min) to 100 (max). A lower score denotes a decline.
Change in Clock Drawing Test (CDT) | 3 months
  The Clock-Drawing Test (CDT) is a simple and effective cognitive test used to assess executive function and visual-spatial function.
  Change is defined as statistical significance in the comparison between before and after the training.
  The score ranges from 0 (min) to 15 (max). A lower score denotes a decline.
Change in Brief Visuospatial Memory Test (BVMT) | 3 months
  The Brief Visuospatial Memory Test (BVMT) measures visuospatial memory.
  Change is defined as statistical significance in the comparison between before and after the training.
  The score ranges from 0 (min) to 36 (max). A lower score denotes a decline.
Change in Symbol Digit Modalities Test (SDMT) | 3 months
  The Symbol Digit Modalities Test (SDMT) is a screening instrument to assess cognitive function and especially processing speed.
  Change is defined as statistical significance in the comparison between before and after the training.
  The score ranges from 0 (min) to 110 (max). Scoring involves summing the number of correct substitutions within the 90-second interval. A lower score denotes a decline.
Change in Verbal Fluency: Phonemic [ Chi-Sigma-Alpha] | 3 months
  Verbal Fluency: Phonemic [ Chi-Sigma-Alpha] is a test of verbal fluency to evaluate the ability to retrieve specific information within restricted search parameters. It can be used as an efficient screening instrument for general verbal functioning.
  Change is defined as statistical significance in the comparison between before and after the training.
  The score ranges from 0 to as many as many different words as possible generated beginning with each of the following three Greek letters: X (Chi), S (Sigma), and A (Alpha) within 60 seconds. A lower score denotes a decline.
Change in Verbal Fluency: Semantic [Animals-Fruits-Objects] | 3 months
  Verbal Fluency: Semantic [Animals-Fruits-Objects] is a test of verbal fluency to evaluate the ability to retrieve specific information within restricted search parameters.
  Change is defined as statistical significance in the comparison between before and after the training.
  The score ranges from 0 to as many as many unique words as possible generated within a semantic category (Animals, Fruits, Objects) in 60 seconds. A lower score denotes a decline.
Change in Digit Span (For-Back-Seq) _WAIS-4GR | 3 months
  Digit Span (For-Back-Seq) _WAIS-4GR is a tool to measure one's verbal short-term and working memory.
  Change is defined as statistical significance in the comparison between before and after the training.
  The score ranges from 0 (min) to 48 (max). A lower score denotes a decline.
Change in Stroop Neuropsychological Test (SNST) | 3 months
  Stroop Neuropsychological Test (SNST) provides a brief screening for brain damage, dysfunction of selective attention, and cognitive flexibility.
  Change is defined as statistical significance in the comparison between before and after the training.
  The score ranges from 0 (min) to the sum of correct answers within 2 minutes. A lower score denotes a decline.
Change in Greek Accentuation Test (GAT) | 3 months
  The Greek Accentuation Test (GAT) is a test of premorbid intellectual functioning.
  Change is defined as statistical significance in the comparison between before and after the training.
  The score ranges from 0 (min) to 50 (max). A lower score denotes a decline.
Change in Depression Anxiety Stress Scale (DASS-21) | 3 months
  Depression Anxiety Stress Scale (DASS-21) is a self-report scale designed to measure the negative emotional states of depression, anxiety, and stress.
  Change is defined as statistical significance in the comparison between before and after the training.
  The score ranges from 0 (min) to 63 (max). A lower score denotes an amelioration or absence of symptoms.
Change in Multiple Sclerosis Impact Scale (MSIS-29) | 3 months
  Multiple sclerosis Impact Scale (MSIS-29) measures coordination, fatigue, flexibility, muscle performance, muscle tone/spasticity, balance/falls, reach and grasp, self-care, health and wellness, leisure, quality of life, role function, social function, and work.
  A 29-item, self-report questionnaire designed to measure the physical and psychological impact of MS.
  Change is defined as statistical significance in the comparison between before and after the training.
  The score ranges from 29 (min) to 116 (max). A lower score denotes an amelioration or absence of symptoms.
Change in the Cognitive Reserve Questionnaire (CRIq) | 3 months
  The Cognitive Reserve Questionnaire (CRIq) is an instrument for measuring cognitive reserve.
  Change is defined as statistical significance in the comparison between before and after the training.
  The questionnaire is divided into 3 sections: CRI-Education, CRI-WorkingActivity, CRI-LeisureTime.
  The CRIq score falls into 1 of 5 ordered levels: low (less than 70); medium-low (70-84); medium (85-114); medium-high (115-130); and high (more than 130). A lower score means a lower cognitive reserve.
Change in Modified Fatigue Impact Scale (MFIS) | 3 months
  The Modified Fatigue Impact Scale (MFIS) is a structured, self-report questionnaire that concerns how fatigue impacts their lives.
  Change is defined as statistical significance in the comparison between before and after the training.
  The score ranges from 0 (min) to 84 (max). A lower score denotes an amelioration or absence of symptoms.
Change in EQ-5D-5L | 3 months
  The EQ-5D-5L is a self-assessed, health-related, quality-of-life questionnaire. The scale measures the quality of life on a 5-component scale including mobility, self-care, usual activities, pain/discomfort, and anxiety/depression.
  Change is defined as statistical significance in the comparison between before and after the training.
  A lower score denotes an amelioration or absence of symptoms.
Change in EQ-5D-5L -EQ-VAS | 3 months
  Change is defined as statistical significance in the comparison between before and after the training.
  The score ranges from 0% (min) to 100% (max). The lower the score, the worse the perception of health.
Change in Beck Depression Inventory-Fast Screen (BDI-FS) | 3 months
  Beck Depression Inventory-Fast Screen (BDI-FS) is a 21-question self-report inventory for measuring the severity of depression.
  Change is defined as statistical significance in the comparison between before and after the training.
  The score ranges from 0 (min) to 21 (max). A lower score denotes an amelioration or absence of symptoms.
Change in Timed 25-Foot Walk (T25-FW) | 3 months
  The Timed 25-Foot Walk (T25-FW) assesses walking speed and general walking ability on a ~8m (7.62m) corridor.
  The T25FW score is calculated by averaging the two tests performed (in seconds).
  Time limit per trial: 3 minutes (180 seconds).
  Change is defined as statistical significance in the comparison between before and after the training.
  An increased measure of timing denotes improvement.
Change in 3 m backwards walk test | 3 months
  The 3 m backwards walk test assesses backward walking which is more sensitive to detecting changes in mobility and balance than walking forward.
  The score records the time (in seconds) per trial.
  Change is defined as statistical significance in the comparison between before and after the training.
  An increased measure of timing denotes improvement.
Change in Hole Peg Test (9-HPT) | 3 months
  The Hole Peg Test (9-HPT) is a brief, standardized, quantitative test that assesses upper extremity functionality, looking at how well the patient can use both their primary and non-primary hand to perform a specific task.
  Time limit per trial: 5 minutes (300 seconds).
  Change is defined as statistical significance in the comparison between before and after the training.
  An increased measure of timing denotes improvement.
Change in Four Square Step Test (FSST) | 3 months
  The Four Square Step Test (FSST) assesses dynamic stability and the subject's ability to step over low objects forward, sideways, and backward.
  The aim is to step as fast as possible into each square with both feet in the following sequence: Square 2, 3, 4, 1, 4, 3, 2, 1 (clockwise to counterclockwise).
  The best time (in seconds) of two FSST is the score.
  Change is defined as statistical significance in the comparison between before and after the training.
  An increased measure of timing denotes improvement.
Change in Single Leg Stance Test (SLS) | 3 months
  The Single Leg Stance Test (SLS): assesses static postural and balance control and is a valuable clinical tool for monitoring neurological and musculoskeletal status as well as for managing fall risk.
  It is tested on both legs.
  Change is defined as statistical significance in the comparison between before and after the training.
  An increased measure of timing denotes improvement.
Change in the Handgrip Strength Test | 3 months
  The Handgrip Strength Test assesses endurance to the maximum strength of the upper limbs. Grip strength is typically measured in kilograms by squeezing a type of muscle strength testing equipment, known as a dynamometer in each hand.
  The average healthy grip strength for men is a squeeze of about 33kg while women typically measure around 20kg.
  Change is defined as statistical significance in the comparison between before and after the training.
  An increased measure of squeeze denotes improvement.

CONTACTS AND LOCATIONS:
Overall Officials: Charis Styliadis, PhD, Principal Investigator — Aristotle University Of Thessaloniki
Locations (1):
- Laboratory of Medical Physics and Digital Innovation, AUTH, Thessaloniki, Central Macedonia, Greece

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Styliadis C, Kartsidis P, Paraskevopoulos E, Ioannides AA, Bamidis PD. Neuroplastic effects of combined computerized physical and cognitive training in elderly individuals at risk for dementia: an eLORETA controlled study on resting states. Neural Plast. 2015;2015:172192. doi: 10.1155/2015/172192. Epub 2015 Apr 7. PMID 25945260
- [Background] Klados MA, Styliadis C, Frantzidis CA, Paraskevopoulos E, Bamidis PD. Beta-Band Functional Connectivity is Reorganized in Mild Cognitive Impairment after Combined Computerized Physical and Cognitive Training. Front Neurosci. 2016 Feb 29;10:55. doi: 10.3389/fnins.2016.00055. eCollection 2016. PMID 26973445
- See also: MS-NEUROPLAST Facebook page — https://www.facebook.com/profile.php?id=100066598856507